CLINICAL TRIAL: NCT00754767
Title: Pilot Study of L-Carnitine Supplementation in the Prevention of Chemotherapy-induced Peripheral Neuropathy in Women With Metastatic Breast Cancer
Brief Title: L-Carnitine L-Tartrate in Preventing Peripheral Neuropathy Caused By Chemotherapy in Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to accrue study participants
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000614311; PNCC-03312-05-C; UMN-0508M72428
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2015-10

CONDITIONS: Breast Cancer; Chemotherapeutic Agent Toxicity; Neurotoxicity
Keywords: neurotoxicity; chemotherapeutic agent toxicity; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neurotoxicity Syndromes | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral L-carnitine L-tartrate twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.
  Interventions: Drug: L-carnitine L-tartrate
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: L-carnitine L-tartrate — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: L-carnitine L-tartrate may prevent peripheral neuropathy caused by chemotherapy.

PURPOSE: This randomized clinical trial is studying how well L-carnitine L-tartrate works in preventing peripheral neuropathy caused by chemotherapy in women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the tolerability and usefulness of the dietary supplement, L-carnitine L-tartrate, in the prevention of chemotherapy-induced peripheral neuropathy in women with metastatic breast cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral L-carnitine L-tartrate twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.
* Arm II: Patients receive oral placebo twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.

Patients complete questionnaires periodically to assess neuropathy, pain, fatigue, sleep, and activities of daily living.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Metastatic disease
* Scheduled to receive ≥ 1 of the following chemotherapy drugs:

  * Paclitaxel
  * Docetaxel
  * Capecitabine
  * Gemcitabine hydrochloride

    * Concurrent enrollment in the University of Minnesota study "Population Pharmacokinetics and Pharmacogenetics of Gemcitabine in Adult Patients with Solid Tumors" (Human Subjects Code 0508M72989) required
  * Albumin-bound paclitaxel (Abraxane)
  * Doxorubicin hydrochloride

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* Serum creatinine < 2.0 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of seizures
* No uncontrolled hypertension
* No history of stroke
* No malabsorption syndrome
* No cognitive impairment
* No history of psychiatric disability affecting informed consent or compliance with drug intake
* Able to take oral medication
* Able to complete questionnaire(s) alone or with assistance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent warfarin
* No concurrent radiotherapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-01-02 (Actual); Primary Completion 2008-04-02 (Actual); Study Completion 2008-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shapiro, PhD, Principal Investigator — Park Nicollet Cancer Center
Locations (2):
- United States (2):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: oncology clinic
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: data was not analyzed due to study termination

OUTCOME MEASURES:

1. Primary Outcome: Vibratory Threshold as Assessed by the Rydel-Seiffer Quantitative Tuning Fork
Description: Data was not analyzed due to study termination
Time Frame: baseline, days 1 and 2 post chemo x 4 cycles
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm I L-Carnitine: Patients receive oral L-carnitine L-tartrate twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.
  L-carnitine L-tartrate: Given orally
- Arm II-Placebo: Patients receive oral placebo twice daily beginning on day 2 of the first course of chemotherapy and continuing until after completion of 4 courses of chemotherapy.
  placebo: Given orally
Arm/Group | Arm I L-Carnitine | Arm II-Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes